CLINICAL TRIAL: NCT00568516
Title: Phase II Study of ASP3550 - A Maintenance-dose Finding Study in Patients With Prostate Cancer
Brief Title: Phase II Study of ASP3550 in Patients With Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3550-CL-0003
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Prostatic Neoplasms
Keywords: ASP3550; Degarelix; Prostate cancer; Prostatic neoplasms
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1.Low dose group (Experimental)
  Interventions: Drug: ASP3550
- 2.High dose group (Experimental)
  Interventions: Drug: ASP3550

INTERVENTIONS:
Drug: ASP3550 — subcutaneous administration
  Other Names: Degarelix

SUMMARY:
To assess the effect of ASP3550 on the maintenance of serum testosterone suppression in patients with prostate cancer

DETAILED DESCRIPTION:
Two doses of ASP3550 were administered to patients with prostate cancer. The primary efficacy variable was the effect of ASP3550 on the maintenance of serum testosterone suppression. In addition, the safety and pharmacokinetics of ASP3550 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Is a male patient with histologically proven prostate cancer (adenocarcinoma) of all stages
* Is a patient in whom endocrine treatment is indicated. Patients with rising serum PSA after having prostatectomy or radiotherapy performed with curative intention may be included
* Has a serum testosterone level above 1.5 ng/mL at screening
* Has an ECOG (Eastern Co-operative Oncology Group) P.S. (Performance Status) score of 0 to 2

Exclusion Criteria:

* Previous or present endocrine treatment for prostate cancer. However, patients who have undergone neoadjuvant/adjuvant endocrine therapy for a maximal duration of 6 months and in whom prostatectomy or radiotherapy was terminated at least 6 months preceding Screening Visit may be included
* Is being treated with a 5α-reductase inhibitor
* Is a candidate for curative therapy, i.e., radical prostatectomy or radiotherapy within 12 months
* Has concurrent or a history of severe asthma (defined as a need for daily treatment with inhalation steroids), anaphylactic reactions, severe urticaria and angioedema

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2007-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with serum testosterone ≤0.5 ng/mL from Day 28 to Day 364 of treatment | 1 Year

SECONDARY OUTCOMES:
Proportion of patients with testosterone surge | 1 Year
Percentage change in serum PSA | 1 Year
Changes in serum levels of testosterone, LH, FSH and PSA over time | 1 Year
Time to the recurrence of serum PSA | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyusyu
  - Shikoku
  - Tōhoku